CLINICAL TRIAL: NCT06091306
Title: Therapeutic Process at Work in Multiple Family Therapy Groups for Anorexia Nervosa During Adolescence. An Exploratory Study.
Brief Title: Qualitative Evaluation of Change Processes in Multifamily Therapy for Adolescents With Anorexia Nervosa
Acronym: QUALI-TMF-TCA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230662; 2023-A00668-37 (Other: ANSM (France))
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Adolescence; Familial relationships; Multiple family therapy groups; Group therapy; Therapeutic process; Qualitative study
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psychotherapy; Psychotherapy, Group

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants in a multifamily therapy group for adolescents, their parents and siblings: The study is therefore being proposed to all the families who have taken part in the multifamily therapy for anorexia nervosa, i.e. the adolescents being followed, their parents and siblings.
  The investigators propose to use a qualitative methodology aimed at collecting the experiences of patients suffering from anorexia nervosa, their parents and their siblings, using alternately, depending on the group, data collection by focus group or by individual semi-structured interview according to a semi-structured interview guide specifically designed by the research team. The data was collected 4 to 6 months after the tenth and final session of the multi-family group.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Multifamily therapy (MFT), which involves bringing several families together to address the problem of anorexia nervosa, has proved effective for several years now.
  Since January 2019, multifamily therapy has been offered to adolescents aged 12 to 18 who are being treated for anorexia nervosa at the Maison de Solenn-Maison des Adolescents at Cochin Hospital, and to their families.
  Each group brings together 5 to 7 families and comprises 10 3-hour sessions, with 3 weeks between each session. 2 groups are offered per year. Multifamily therapy therefore involves 10 to 14 families per year. It complements the other approaches available in the department.
  Other Names: Multifamily Therapy for anorexia nervosa during adolescence

SUMMARY:
Anorexia nervosa is a characterised disorder which forms part of the wider spectrum of eating disorders. It is a common pathology, particularly in adolescence, with a complex, severe prognosis in both somatic and psychiatric terms, and significant psychosocial consequences, particularly for family relationships.

The treatment of anorexia requires a multidisciplinary team of specialists who can offer individual and family-based approaches. International recommendations highlight the encouraging results of family therapy in the treatment of anorexia nervosa in adolescence. Various types of family approach exist, including "Family Based Treatments", which are a specific but highly effective approach, particularly widespread in the United States. Multifamily therapy (MFT), which involves bringing several families together to address the problem of anorexia, has proved effective for several years now.

Since January 2019, multifamily therapy has been offered to adolescents aged 12 to 18 who are being followed at the Maison de Solenn-Maison des Adolescents at Cochin hospital, for anorexia nervosa, as well as their families.

Each group brings together 5 to 7 families and comprises 10 3-hour sessions, with 3 weeks between each session. 2 groups are offered per year. Multi-family therapy therefore involves 10 to 14 families per year. It complements the other approaches available in the department.

To be able to describe the therapeutic processes at work in multifamily groups in order to be able to better describe our therapeutic device and envisage possible modifications. These processes would be broken down into four areas: MFT and its effects on the anorexic symptom, MFT and its effects on the family, MFT as group therapy and ways of improving the MFT system.

DETAILED DESCRIPTION:
Anorexia nervosa is a characterised disorder which forms part of the wider spectrum of eating disorders. It is a common pathology, particularly in adolescence, with a complex, severe prognosis in both somatic and psychiatric terms, and significant psychosocial consequences, particularly for family relationships.

The treatment of anorexia requires a multidisciplinary team of specialists who can offer individual and family-based approaches. International recommendations highlight the encouraging results of family therapy in the treatment of anorexia nervosa. Various types of family approach exist, including "Family Based Treatments", which are a specific but highly effective approach, particularly widespread in the United States. Multifamily therapy (MFT), which involves bringing several families together to address the problem of anorexia, has proved effective for several years now.

Since January 2019, multifamily therapy has been offered to adolescents aged 12 to 18 who are being followed at the Maison de Solenn-Maison des Adolescents at Cochin Hospital for anorexia nervosa, as well as their families.

Each group brings together 5 to 7 families and comprises 10 3-hour sessions, with 3 weeks between each session. 2 groups are offered per year. Multi-family therapy therefore involves 10 to 14 families per year. It complements the other approaches available in the department.

Primary objective:

To be able to describe the therapeutic processes at work in these multifamily groups in order to be able to better describe our therapeutic device and envisage possible modifications. These processes would be broken down into four areas: MFT and its effects on the anorexic symptom, MFT and its effects on the family, MFT as a group therapy and ways of improving the MFT system.

Secondary objectives:

* MFT and its effect on the symptom: to better describe and analyse the processes at work in multifamily therapy that lead to symptomatic improvement in adolescents through the perception of the adolescent himself, his parents or his brothers and sisters.
* MFT and its effects on the family: to describe in detail the psychotherapeutic processes within the MFT system that are involved in changing family relationships.
* MFT and its effects as group therapy: The context of group therapy is often a powerful lever/motivator of change and the investigators are seeking to better describe and understand the mechanisms at play in the group and how this influences the family and the anorexic symptom.
* Areas for improvement in MFT: Our study also aims to determine, in the context of a multifamily group for anorexia nervosa, the therapeutic contexts (single-family, intragenerational, multigenerational) and therapeutic mediations most conducive to change, in order to improve our practice and therapeutic proposals.

The study is therefore being proposed to all the families who have taken part in the multifamily therapy for anorexia nervosa, i.e. the adolescents being followed, their parents and siblings.

The investigators propose to use a qualitative methodology aimed at collecting the experiences of patients suffering from anorexia nervosa, their parents and their siblings, using alternately, depending on the group, data collection by focus group or by individual semi-structured interview according to a semi-structured interview guide specifically designed by the research team. The data was collected 4 to 6 months after the tenth and final session of the multifamily group.

The theoretical framework is qualitative and no statistical comparison is expected.

The investigators chose to use Interpretative Phenomenological Analysis (IPA) to study the meaning that the subject constructs from lived experiences. IPA is a recognised method of content analysis, particularly in health psychology.

Approximately 3 months after the end of a multifamily group on anorexia nervosa, the investigators will contact the families by telephone or e-mail to invite the families to take part in research interviews which will take place 4 to 6 months after the tenth and last session of the multifamily group in which the family took part.

The investigators will arrange to meet the families in the department on the same day to carry out an information interview, collect non-oppositions, interviews to collect socio-demographic data and then individual semi-structured interviews or focus groups (depending on staff availability).

The qualitative analysis of our research concerns the thematic analysis of the participants' discourse (adolescent patients, parents and siblings of these adolescents), so the main evaluation criterion concerns the extraction of sufficiently rich material from the discourse to carry out this analysis.

ELIGIBILITY:
Inclusion Criteria:

Families who have taken part in a multifamily group on anorexia nervosa, i.e. :

* Parents (or any adult identified as a referent by the teenager), teenagers and siblings (over 6 years old) who have taken part in multi-family therapy (people from the teenager's family who have not taken part in the group will not be included),
* Adolescents aged 12 to 20,
* Adolescents with anorexia nervosa according to DSM5 criteria,
* Adolescents treated at the Maison des Adolescents at Cochin Hospital,
* Non-opposition of adolescents, their parents and siblings.

It will be possible to include in the study a parent or sibling whose adolescent did not wish to take part in the research but who participated in the MFT group.

Exclusion Criteria:

* Contraindication to multifamily therapy (i.e. any family situation that makes it impossible to bring parents and children together in family therapy without changing the setting (parents stripped of parental authority, educational removal measure, mediated visits, etc.),
* Any patient whose main diagnosis is not anorexia nervosa according to DSM5 criteria.
* Patients with an autistic spectrum disorder, a chronic psychotic disorder or an intellectual disability as their primary or secondary diagnosis according to DSM 5.
* Participants under curatorship or guardianship
* Participants not covered by a Social Security scheme.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study is therefore being offered to all families who have taken part in multifamily therapy for anorexia nervosa, i.e. the adolescent patients being treated for anorexia nervosa, their parents and siblings.
  These patients and their families come from the clinical population followed in our institution for anorexia nervosa: the Maison des Adolescents of the Cochin Hospital - Maison de Solenn (APHP, Paris). Participation in a multi-family group is complementary to the usual care provided in the department (psychiatric, pediatric and dietetic follow-up) and does not replace the usual individual care.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Semi-structured qualitative interviews | Day of inclusion
  Semi-structured individual or group (focus group) interviews following a pre-designed interview guide.
  The qualitative analysis of our research concerns the thematic analysis of the participants' discourse (adolescent patients, parents and siblings of these adolescents), so the main evaluation criterion concerns the extraction of sufficiently rich material from the discourse to carry out this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Rose MORO, MD, PhD, Study Director — University Hospital Cochin, Maison des Adolescents - Youth Department, F-75014 Paris, France; Salomé Grandclerc, MD, Principal Investigator — University Hospital Cochin, Maison des Adolescents - Youth Department, F-75014 Paris, France
Locations (1):
- University Hospital Cochin, Maison des Adolescents - Youth Department (Maison de Solenn), Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No